CLINICAL TRIAL: NCT00000496
Title: Platelet Drug Trial in Coronary Disease Progression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 15
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2012-04

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia | interventions — Aspirin; Dipyridamole

INTERVENTIONS:
Drug: aspirin
Drug: dipyridamole

SUMMARY:
To determine the effectiveness of the platelet inhibitor drugs dipyridamole and aspirin in reducing the angiographic progression of coronary artery disease over a five-year period and to test the predictive value of the platelet survival half-life in identifying patients with more rapid progression of coronary disease and development of its complications.

DETAILED DESCRIPTION:
BACKGROUND:

Coronary atherosclerosis is the leading cause of death in this country and the developed countries of the world. Although modern coronary care units have resulted in a markedly decreased hospital mortality from acute myocardial infarction, especially in those patients who enter the hospital early, its overall impact is limited since two-thirds of patients who die from coronary disease do not reach the hospital. When the trial was initiated in 1979, new approaches to the medical treatment of coronary disease and its complications were needed with an effort directed towards prevention of its progression and prevention of its complications through medical therapy. This prevention could save significant health care dollars over the long-term especially if the need for aortocoronary bypass graft surgery and the incidence of myocardial infarction could be reduced. Early identification of the patient at risk of developing coronary disease or of those with early coronary artery lesions would allow a greater impact of any successful intervention therapy.

DESIGN NARRATIVE:

Randomized, double-blind. The patients in the experimental group were treated with dipyridamole and aspirin for five years. Patients in the control group received a lactose placebo. The primary endpoint was angiographic evidence of progression of coronary artery disease and development of new coronary disease. Secondary endpoints included total mortality, cardiac mortality, mortality due to myocardial infarction, and incidence of new myocardial infarction. Recruitment ended in December 1982.

The study completion date listed in this record was obtained from the statement immediately above ("Recruitment ended in December 1982") and was confirmed from the Query/View/Report (QVR) System.

ELIGIBILITY:
Patients aged 65 or less. Angiographically identified coronary heart disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1979-12; Study Completion 1982-12 (Actual)